CLINICAL TRIAL: NCT02881554
Title: Functional Liver Imaging With Sulfur Colloid SPECT/CT in Primary and Metastatic Liver Cancer Patients Receiving Liver-Directed Treatment: A Pilot Study
Brief Title: Sulfur Colloid SPECT/CT in Measuring Liver Function in Patients With Primary or Metastatic Liver Cancer Undergoing Radiation Therapy or Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to low accrual in Cohort B. (Accrual goal for Cohort A was met.)
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Smith Apisarnthanarax, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9646; NCI-2016-01198 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9646 (Other: Fred Hutch/University of Washington Cancer Consortium); RG3116003 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2016-08-23; First posted 2016-08-29 (Estimated); Results first posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma; Intrahepatic Cholangiocarcinoma; Stage IV Liver Cancer; Stage IVA Liver Cancer; Stage IVB Liver Cancer; Vascular Thrombosis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Liver Neoplasms; Thrombosis | interventions — X-Rays; Photons; Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (SC SPECT/CT) (Experimental): There are 2 cohorts of patients: Those receiving radiation therapy per standard of care (Cohort A) and those undergoing surgery per standard of care (Cohort B). All patients have a total of 3 SPECT/CT imaging with 99mTc-SC. The first scan in both cohorts is routine medical care (not experimental) and takes place prior to initiation of RT or surgery. Two follow up scans are part of the protocol.
  * In cohort A, the first follow up scan occurs at mid-RT, and the second one at 1 month post-RT.
  * In cohort B, the first follow-up scan occurs 3-5 days postoperatively, and the second one at 1 month post-operatively. An additional IV contrast enhanced CT scan (70 second delay) will be obtained immediately following the SPECT/CT scan for all 3 SPECT/CT scans.
  Interventions: Procedure: Computed Tomography; Procedure: Single Photon Emission Computed Tomography; Drug: Technetium Tc-99m Sulfur Colloid

INTERVENTIONS:
Procedure: Computed Tomography — Undergo SC SPECT/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT SCAN; tomography
Procedure: Single Photon Emission Computed Tomography — Undergo SC SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Drug: Technetium Tc-99m Sulfur Colloid — Given IV
  Other Names: Tc 99m Sulfur Colloid; Tc-99m SC; Technetium Tc 99m Sulfur Colloid

SUMMARY:
This pilot trial studies how well single photon emission computed tomography (SPECT)/computed tomography (CT) with technetium Tc-99m sulfur colloid works in measuring liver function in patients with liver cancer that has or has not spread to other place in the body who are undergoing radiation therapy or surgery. Diagnostic procedures, such as sulfur colloid SPECT/CT scans, may measure normal liver tissue before, during and after treatment and help doctors plan better treatment for liver cancer patients.

DETAILED DESCRIPTION:
OUTLINE: Patients are assigned to 1 of 2 cohorts depending on which standard of care they are receiving outside of this study, as part of their cancer treatment: radiation treatment (RT) or surgery.

All patients have a total of 3 SPECT/CT imaging with 99mTc-SC. The first scan in both cohorts is routine medical care (not experimental) and takes place prior to initiation of RT or surgery. Two follow up scans are part of the protocol.

COHORT A (patients receiving radiation therapy per standard cancer treatment): The first follow up scan occurs at mid-RT, and the second one at 1 month post-RT.

COHORT B (patients undergoing surgery per standard cancer treatment): The first follow-up scan occurs 3-5 days postoperatively, and the second one at 1 month post-operatively. An additional intravenous (IV) contrast enhanced CT scan (70 second delay) will be obtained immediately following the SPECT/CT scan for all 3 SPECT/CT scans.

After completion of study, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of hepatocellular carcinoma (HCC), intrahepatic cholangiocarcinoma, or metastatic liver cancer planned to receive definitive doses of radiation or surgical resection are eligible
* Measurable hepatic disease and/or presence of vascular tumor thrombosis
* Diagnostic CT or magnetic resonance imaging (MRI) scan within 2 months of study entry
* There are no limits on prior therapy; patients are allowed to have prior systemic therapy, radiation therapy, radiofrequency ablation, catheter-based therapies, and surgery; patients are allowed to have concurrent chemotherapy with radiation treatment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients unable to tolerate a SPECT/CT 99mTc-SC scan
* Patients who are not planning to adhere to the required follow up schedule as outlined in this protocol
* Pregnant women
* Women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception
* Patients unable to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Smith Apisarnthanarax, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - ProCure Proton Therapy Center-Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SC SPECT/CT: Cohort A - Radiation: Cohort A includes all subjects receiving radiation therapy per standard of care. Patients have a total of 3 SPECT/CT imaging with 99mTc-SC. The first scan in both cohorts is routine medical care (not experimental) and takes place prior to initiation of radiation treatment (RT) or surgery. Two follow up scans are part of the protocol.
  The first follow up scan occurs at mid-RT, and the second one at 1-month post-RT.
  Computed Tomography: Undergo SC SPECT/CT
  Single Photon Emission Computed Tomography: Undergo SC SPECT/CT
  Technetium Tc-99m Sulfur Colloid: Given IV
- SC SPECT/CT: Cohort B - Surgery: Cohort B includes all subjects undergoing surgery per standard of care. Patients have a total of 3 SPECT/CT imaging with 99mTc-SC. The first scan in both cohorts is routine medical care (not experimental) and takes place prior to initiation of RT or surgery. Two follow up scans are part of the protocol.
  The first follow-up scan occurs 3-5 days postoperatively, and the second one at 1 month post-operatively. An additional IV contrast enhanced CT scan (70 second delay) will be obtained immediately following the SPECT/CT scan for all 3 SPECT/CT scans.
  Computed Tomography: Undergo SC SPECT/CT
  Single Photon Emission Computed Tomography: Undergo SC SPECT/CT
  Technetium Tc-99m Sulfur Colloid: Given IV
Period: Overall Study
Arm/Group | SC SPECT/CT: Cohort A - Radiation | SC SPECT/CT: Cohort B - Surgery
Started | 38 | 3
Completed | 36 | 3
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- SC SPECT/CT: Cohort A - Radiation: Cohort A includes all subjects receiving radiation therapy per standard of care. Patients have a total of 3 SPECT/CT imaging with 99mTc-SC. The first scan in both cohorts is routine medical care (not experimental) and takes place prior to initiation of RT or surgery. Two follow up scans are part of the protocol.
  The first follow up scan occurs at mid-RT, and the second one at 1-month post-RT.
  Computed Tomography: Undergo SC SPECT/CT
  Single Photon Emission Computed Tomography: Undergo SC SPECT/CT
  Technetium Tc-99m Sulfur Colloid: Given IV
- Total: Total of all reporting groups
Arm/Group | SC SPECT/CT: Cohort A - Radiation | SC SPECT/CT: Cohort B - Surgery | Total
Number analyzed (Participants) | 38 | 3 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 1 | 8
  >=65 years | 31 | 2 | 33
Age, Continuous [Mean (Full Range); unit: years] | 71.87 [29 to 96] | 74.67 [64 to 80] | 72.07 [29 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 1 | 16
  Male | 23 | 2 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 34 | 3 | 37
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 38 | 3 | 41

OUTCOME MEASURES:

1. Primary Outcome: Longitudinal Changes in Liver Function as Measured by SC SPECT/CT Functional Liver Volume: Cohort A - Radiation
Description: Functional liver volume ratio (FLV): represents the percent of the anatomic liver which is functioning and is defined as the ratio of liver functional volume (in cc of volume) to the anatomic liver volume (in cc of volume). Since this outcome measure is a ratio, it is unitless. A higher FLV ratio reflects a higher volume of functional liver.
Time Frame: Baseline, mid-treatment at 2 weeks, and post-treatment at 1 month
Population: Only participants in Cohort A with evaluable treatment scans were assessed for this outcome.
Measure: Median (Full Range); unit: ratio
Arm/Group | SC SPECT/CT: Cohort A - Radiation
Number analyzed (Participants) | 36
ratio
  Baseline FLV Ratio | 0.36 [0.01 to 0.63]
  Mid-Treatment FLV Ratio | 0.34 [0.00 to 0.67]
  Post-Treatment FLV Ratio | 0.25 [0.00 to 0.58]

2. Primary Outcome: Longitudinal Changes in Liver Function as Measured by SC SPECT/CT Liver-to-Spleen Mean: Cohort A - Radiation
Description: Liver-to-spleen ratio (L/S mean): represents the magnitude of the global liver function and is defined as the ratio of the mean SC counts in the functional liver to the mean SC counts in the spleen. Since this outcome measure is a ratio, it is unitless. A higher L/S mean ratio reflects higher magnitude of liver function.
Time Frame: Baseline, mid-treatment at 2 weeks, and post-treatment at 1 month
Population: Only participants in Cohort A with evaluable treatment scans were assessed for this outcome.
Measure: Median (Full Range); unit: ratio
Arm/Group | SC SPECT/CT: Cohort A - Radiation
Number analyzed (Participants) | 36
ratio
  Baseline L/S Ratio | 1.11 [0.37 to 2.83]
  Mid-Treatment L/S Ratio | 0.96 [0.38 to 2.83]
  Post-Treatment L/S Ratio | 0.71 [0.22 to 2.76]

3. Primary Outcome: Longitudinal Changes in Liver Function as Measured by SC SPECT/CT Total Liver Function: Cohort A - Radiation
Description: Total liver function (TLF): represents the integral liver function and is defined by the product of the functional liver volume (FLV) ratio and liver-to-spleen (L/S) mean ratio. Since this outcome measure is a product of ratios, it is unitless. A higher TLF ratio reflects higher liver function. Median differences were estimated using Wilcoxon (Mann-Whitney) tests.
Time Frame: Baseline, mid-treatment at 2 weeks, and post-treatment at 1 month
Population: Only participants in Cohort A with evaluable treatment scans were assessed for this outcome.
Measure: Median (Full Range); unit: ratio
Groups:
- All Patients: Includes all subjects who received 3 SPECT/CT imaging with 99mTc-SC: baseline, mid-treatment, and post-treatment.
- Child-Pugh A Patients: Sub-population of patients with Child-Pugh A liver function who received 3 SPECT/CT imaging with 99mTc-SC: baseline, mid-treatment, and post-treatment.
- Child-Pugh B/C Patients: Sub-population of patients with Child-Pugh B and C liver function who received 3 SPECT/CT imaging with 99mTc-SC: baseline, mid-treatment, and post-treatment.
Arm/Group | All Patients | Child-Pugh A Patients | Child-Pugh B/C Patients
Number analyzed (Participants) | 36 | 22 | 11
ratio
  Baseline TLF Ratio | 0.41 [0.00 to 1.78] | 0.44 [0.05 to 1.78] | 0.18 [0.00 to 0.55]
  Mid-Treatment TLF Ratio | 0.29 [0.00 to 1.29] | 0.39 [0.11 to 1.29] | 0.15 [0.00 to 0.72]
  Post-Treatment TLF Ratio | 0.18 [0.00 to 1.60] | 0.29 [0.03 to 1.60] | 0.09 [0.00 to 0.38]
Statistical Analysis 1: Comparison: All Patients; Null hypothesis = no difference in TLF between mid-treatment and baseline. Wilcoxon (Mann-Whitney) tests were performed assessing the longitudinal difference between mid-treatment TLF from baseline TLF; Test type: Other — Non-parametric; p < 0.05, Wilcoxon (Mann-Whitney) — Statistically significant p-value is <0.05; Median Difference (Final Values) = 0.12
Statistical Analysis 2: Comparison: All Patients; Null hypothesis = no difference in TLF between mid-treatment and baseline. Wilcoxon (Mann-Whitney) tests were performed assessing the longitudinal difference between post-treatment TLF from baseline TLF; Test type: Other — Non-parametric; p < 0.001, Wilcoxon (Mann-Whitney) — Statistically significant p-value is <0.05; Median Difference (Final Values) = 0.23
Statistical Analysis 3: Comparison: Child-Pugh A Patients; [analysis description as in outcome 3, analysis 1]; Test type: Other — Non-parametric; p < 0.05, Wilcoxon (Mann-Whitney) — Statistically significant p-value is <0.05; Median Difference (Final Values) = 0.05
Statistical Analysis 4: Comparison: Child-Pugh A Patients vs Child-Pugh B/C Patients; [analysis description as in outcome 3, analysis 2]; Test type: Other — Non-parametric; p < 0.01, Wilcoxon (Mann-Whitney) — Statistically significant p-value is <0.05; Median Difference (Final Values) = 0.15
Statistical Analysis 5: Comparison: Child-Pugh B/C Patients; [analysis description as in outcome 3, analysis 1]; Test type: Other — Non-parametric; p = 0.13, Wilcoxon (Mann-Whitney) — Statistically significant p-value is <0.05; Median Difference (Final Values) = 0.03
Statistical Analysis 6: Comparison: Child-Pugh B/C Patients; [analysis description as in outcome 3, analysis 2]; Test type: Other — Non-parametric; p < 0.05, Wilcoxon (Mann-Whitney) — Statistically significant p-value is <0.05; Median Difference (Final Values) = 0.09
Statistical Analysis 7: Comparison: Child-Pugh A Patients; Null hypothesis = no monotonic association between the baseline TLF and Child-Pugh scores. Spearman rank correlation was performed to assess association between baseline TLF and Child-Pugh scores; Test type: Other — Non-parametric; p = 0.002, Spearman rank correlation — Statistically significant p-value is <0.05; Spearman's correlation coefficient = -0.61

4. Primary Outcome: Longitudinal Changes in Liver Function as Measured by SC SPECT/CT Spatial Heterogeneity: Cohort A - Radiation
Description: To characterize spatial distribution of functional liver, the coefficient of variation (CV) within the FLV will be measured (unitless). A higher CV means more variability or heterogeneity in liver function.
Time Frame: Baseline, mid-treatment at 2 weeks, and post-treatment at 1 month
Population: Only participants in Cohort A with evaluable treatment scans were assessed for this outcome.
Measure: Median (Full Range); unit: ratio
Arm/Group | SC SPECT/CT: Cohort A - Radiation
Number analyzed (Participants) | 36
ratio
  Baseline CV Ratio | 0.38 [0.28 to 0.69]
  Mid-Treatment CV Ratio | 0.40 [0.29 to 0.89]
  Post-Treatment CV Ratio | 0.54 [0.35 to 0.84]

5. Secondary Outcome: Longitudinal Changes in Liver Function as Measured by SC SPECT/CT Functional Liver Volume: Cohort B - Surgery
Description: as for outcome 1
Time Frame: Baseline, perioperative (2-3 days post surgery), and postoperative (1 month post surgery)
Population: Cohort B - Only patients undergoing surgery
Measure: Median (Full Range); unit: ratio
Arm/Group | SC SPECT/CT: Cohort B - Surgery
Number analyzed (Participants) | 3
ratio
  Preoperative FLV Ratio | 0.52 [0.39 to 0.58]
  Perioperative FLV Ratio | 0.59 [0.52 to 0.67]
  Postoperative FLV Ratio | 0.54 [0.53 to 0.64]

6. Secondary Outcome: Longitudinal Changes in Liver Function as Measured by SC SPECT/CT Liver-to-Spleen Mean: Cohort B - Surgery
Description: as for outcome 2
Time Frame: Baseline, perioperative (2-3 days post surgery), and postoperative (1 month post surgery)
Population: Cohort B - Only patients undergoing surgery
Measure: Median (Full Range); unit: ratio
Arm/Group | SC SPECT/CT: Cohort B - Surgery
Number analyzed (Participants) | 3
ratio
  Preoperative L/S Ratio | 1.53 [1.48 to 2.08]
  Perioperative L/S Ratio | 1.23 [1.10 to 2.78]
  Postoperative L/S Ratio | 1.71 [0.91 to 2.57]

7. Secondary Outcome: Longitudinal Changes in Liver Function as Measured by SC SPECT/CT Total Liver Function: Cohort B - Surgery
Description: as for outcome 3
Time Frame: Baseline, perioperative (2-3 days post surgery), and postoperative (1 month post surgery)
Population: Cohort B - Only patients undergoing surgery
Measure: Median (Full Range); unit: ratio
Arm/Group | SC SPECT/CT: Cohort B - Surgery
Number analyzed (Participants) | 3
ratio
  Preoperative TLF Ratio | 0.89 [0.57 to 1.09]
  Perioperative TLF Ratio | 0.73 [0.64 to 1.63]
  Postoperative TLF Ratio | 1.1 [0.49 to 1.37]

ADVERSE EVENTS:
Time Frame: Serious and Other AEs and All-Cause Mortality were assessed for up to 5 years.
Arm/Group | SC SPECT/CT: Cohort A - Radiation | SC SPECT/CT: Cohort B - Surgery
All-Cause Mortality (participants affected / at risk) | 22/36 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/3
Other Adverse Events (participants affected / at risk) | 0/36 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT02881554/Prot_SAP_000.pdf